CLINICAL TRIAL: NCT05009992
Title: A Combination Therapy Trial Using an Adaptive Platform Design for Children and Young Adults With Diffuse Midline Gliomas (DMGs) Including Diffuse Intrinsic Pontine Gliomas (DIPGs) at Initial Diagnosis, Post-Radiation Therapy and at Time of Progression
Brief Title: Combination Therapy for the Treatment of Diffuse Midline Gliomas
Acronym: PNOC022
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: The Chad-Tough Defeat DIPG Foundation (Unknown); Mithil Prasad Foundation (Unknown); Storm the Heavens Fund (Unknown); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Jazz Pharmaceuticals (Industry); Neeve Kolte and Brave Ronil Foundation (Unknown); Will Meeker Foundation (Unknown); CV Biomanufacturing (Unknown)
Responsible Party: Principal Investigator, Sabine Mueller, MD, PhD, Principal Investigator, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200821; NCI-2021-08386 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); 1R01NS124607-01 (NIH)
Record Dates: First submitted 2021-08-10; First posted 2021-08-18 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Intrinsic Pontine Glioma; Diffuse Midline Glioma, H3 K27M-Mutant; Recurrent Diffuse Intrinsic Pontine Glioma; Recurrent Diffuse Midline Glioma, H3 K27M-Mutant; Recurrent WHO Grade III Glioma; WHO Grade III Glioma
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma | interventions — TIC10 compound; Radiotherapy; Phosphatidylinositol 3-Kinases; Proto-Oncogene Proteins c-akt; GDC-0084

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- NOT CURRENTLY ENROLLING - ARM 2: ONC201 (Day -1), Radiation+ONC201, Paxalisib+ONC201 (Experimental): Participants may receive a safety lead in of ONC201. During the trial validation phase, participants without prior biopsy receive ONC201 PO on day -1 prior to standard of care biopsy. During the radiation/re-irradiation phase, participants without prior radiation therapy or have disease progression after radiation therapy undergo weekly radiation therapy and receive ONC201 PO weekly during radiation therapy. During the maintenance phase, participants receive ONC201 PO weekly and paxalisib PO daily (QD). Cycles repeat every 28 days (4 weeks) in the absence of adverse events of unacceptable toxicity
  Interventions: Drug: ONC201; Radiation: Radiation Therapy; Drug: Paxalisib
- NOT CURRENTLY ENROLLING - ARM 4: ONC201 (Day -1,-2), Radiation+ONC201, Paxalisib+ONC201 (Experimental): Participants may receive a safety lead in of ONC201. During the trial validation phase, participants without prior biopsy receive ONC201 PO on days -2 and -1 prior to standard of care biopsy. During the radiation/re-irradiation phase, participants may receive ONC201 PO weekly during radiation therapy. During the maintenance phase, participants receive ONC201 PO weekly and paxalisib PO QD. Cycles repeat every 28 days (4 weeks) in the absence of adverse events or unacceptable toxicity
  Interventions: Drug: ONC201; Radiation: Radiation Therapy; Drug: Paxalisib
- NOT CURRENTLY ENROLLING - ARM 6: Paxalisib (Day -1), Radiation+Paxalisib , Paxalisib+ONC201 (Experimental): Participants may receive a safety lead in of ONC201. During trial validation phase, participants without prior biopsy receive paxalisib PO on day -1 prior to standard of care biopsy. During the radiation/re-irradiation phase, participants without prior radiation therapy or have disease progression after radiation therapy undergo weekly radiation therapy and receive paxalisib PO daily during radiation therapy. During the maintenance phase, participants receive ONC201 PO weekly and paxalisib PO QD. Cycles repeat every 28 days (4 weeks) in the absence of adverse events of unacceptable toxicity
  Interventions: Drug: ONC201; Radiation: Radiation Therapy; Drug: Paxalisib
- Cohort 4 - Dose Escalation, Starting Dose 2 (625mg ONC201) (Experimental): Participants will receive a safety lead in of 625mg (or weight-adjusted adult equivalent RP2D for pediatrics) of ONC201 on Day 1 and 2 of each week. During the target validation phase, participants without prior biopsy receive ONC201 PO on days -2 and -1 prior to standard of care biopsy. For participants receiving non-interventional radiation/re-irradiation per standard of care treatment, participants will receive 625 mg as the starting dose of ONC201 Days 1 and 2 on a weekly basis during radiation. Cycles repeat every 28 days (4 weeks) in the absence of adverse events or unacceptable toxicity
  Interventions: Drug: ONC201; Radiation: Radiation Therapy
- Cohort 5 - ONC201 + Targeted therapies (Experimental): Participants will receive a starting dose of 625mg (or weight-adjusted adult equivalent RP2D for pediatrics) of ONC201 on Day 1 and 2 of each week in combination with targeted agents to be selected from approved/available agents based on a rational therapy approach guided by molecular data from the tumor tissue or cerebral spinal fluid (CSF). For participants receiving non-interventional radiation/re-irradiation per standard of care treatment, prior to starting the combination therapy, participants will receive 625 mg as the starting dose of ONC201 Days 1 and 2 on a weekly basis during radiation. Observations and schedule of events will be issued based on the chosen agent determined to best fit the molecular profile (e.g. BRAFV600E, PDGFRA, FGFR1, NF1).
  Interventions: Drug: ONC201; Radiation: Radiation Therapy
- Cohort 6 - DNX-2401 Repeated Intratumoral Administration (Experimental): Participants will receive repeated DNX-2401 intratumoral infusions every 30 days, for a maximum of six injections. During Infusion 1 and Infusion 3, participants will have a biopsy for tumor tissue collection.
  Interventions: Drug: DNX-2401

INTERVENTIONS:
Drug: ONC201 — Given orally (PO)
  Other Names: TIC10; Antagonist of dopamine receptor D2 (DRD2) and caseinolytic protease proteolytic subunit (ClpP)
  Arms: Cohort 4 - Dose Escalation, Starting Dose 2 (625mg ONC201); Cohort 5 - ONC201 + Targeted therapies; NOT CURRENTLY ENROLLING - ARM 2: ONC201 (Day -1), Radiation+ONC201, Paxalisib+ONC201; NOT CURRENTLY ENROLLING - ARM 4: ONC201 (Day -1,-2), Radiation+ONC201, Paxalisib+ONC201; NOT CURRENTLY ENROLLING - ARM 6: Paxalisib (Day -1), Radiation+Paxalisib , Paxalisib+ONC201
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Radiotherapy
  Arms: Cohort 4 - Dose Escalation, Starting Dose 2 (625mg ONC201); Cohort 5 - ONC201 + Targeted therapies; NOT CURRENTLY ENROLLING - ARM 2: ONC201 (Day -1), Radiation+ONC201, Paxalisib+ONC201; NOT CURRENTLY ENROLLING - ARM 4: ONC201 (Day -1,-2), Radiation+ONC201, Paxalisib+ONC201; NOT CURRENTLY ENROLLING - ARM 6: Paxalisib (Day -1), Radiation+Paxalisib , Paxalisib+ONC201
Drug: Paxalisib — Given PO
  Other Names: Inhibitor of the phosphatidylinositol 3-kinase (PI3K) /Protein kinase B (AKT)/Mechanistic target of rapamycin (mTOR) pathway; GDC-0084; GDC0084; PI3K Inhibitor GDC-0084
  Arms: NOT CURRENTLY ENROLLING - ARM 2: ONC201 (Day -1), Radiation+ONC201, Paxalisib+ONC201; NOT CURRENTLY ENROLLING - ARM 4: ONC201 (Day -1,-2), Radiation+ONC201, Paxalisib+ONC201; NOT CURRENTLY ENROLLING - ARM 6: Paxalisib (Day -1), Radiation+Paxalisib , Paxalisib+ONC201
Drug: DNX-2401 — DNX-2401 is an oncolytic adenovirus that will be administered through direct intratumoral infusion of DNX-2401 via a specialized Neuro Ventricular Cannula.
  Arms: Cohort 6 - DNX-2401 Repeated Intratumoral Administration

SUMMARY:
This phase II trial determines if the combination of ONC201 with different drugs is effective for treating participants with diffuse midline gliomas (DMGs). Despite years of research, little to no progress has been made to improve outcomes for participants with DMGs, and there are few treatment options. This trial will utilize an adaptive platform design in that the different treatment arms for each cohort will be opened and closed based on ongoing preclinical investigation as well as evolving outcome data from the trial.

Novel agents will be continuously added to this study as pre-clinical data emerge to suggest additive or synergistic activity when combined ONC201. Should a novel agent not have an RP2D at the time of incorporation into this study, a phase 1 lead-in will be performed prior to initiation of combination therapy (via study amendment).

DETAILED DESCRIPTION:
OUTLINE:

This is a multi-arm/cohort, multi-institutional, open-label trial. The study is divided into cohorts based on stage of disease (newly-diagnosed, post-radiation therapy without disease progression, and at disease progression).

---THIS STUDY IS NOT ENROLLING ON COHORTS 1, 2, AND 3 --

ENROLLING:

* Cohort 4: Participants in Cohort 4 will be treated with escalating doses of ONC201 based on evolving pharmacokinetic (PK) data available for ONC201.
* Cohort 5: Participants in Cohort 5 will be treated with escalating doses of ONC201 based on evolving PK data and in combination with targeted therapy (or therapies determined by tumor molecular sequencing).
* Cohort 6: Participants in cohort 6 will be treated with repeated intratumoral injections of DNX-2401.

PRIMARY OBJECTIVES:

I. To assess efficacy of combination therapy with ONC201 (ONC201) and novel agent in participants with DMG based on median progression-free survival at 6 months (PFS6) (Cohorts 1 and 2).

II. To assess efficacy of combination therapy with ONC201 and novel agent in participants with recurrent DMG based on overall survival at 7 months (OS7) (Cohort 3).

III. To assess the safety and toxicity of a revised ONC201 dose and dosing schedule in participants with DMG. (Cohort 4).

IV. To assess the safety and toxicity of a revised ONC201 dosing schedule in combination with radiation or re-irradiation in participants with DMG. (Cohort 4).

V. To evaluate the pharmacokinetic profile of a revised ONC201 dose and dosing schedule in participants with DMG. (Cohort 4).

VI. To assess the safety and toxicity of ONC201 with agent(s) that will be determined by a specialized tumor board recommendation that is based on molecular assessments of tumor tissue or cerebrospinal fluid (CSF). (Cohort 5).

VII. To determine the maximum tolerated number of intratumor infusions of DNX-2401, with a maximum of 6, in participants with thalamic or pontine DMG who completed radiotherapy. (Cohort 6, Phase 1) VIII. To assess efficacy of repeated intratumor infusions with DNX-2401 in participants with DMG based on overall survival at 15 months. (Cohort 6, expansion cohort)

EXPLORATORY OBJECTIVES:

I. To confirm blood brain barrier (BBB) penetration of ONC201 in DMGs by measuring the concentration of ONC201 in tumor tissue (All cohorts except Cohort 6; target validation phase).

II. To confirm BBB penetration of novel agents in DMGs by measuring the concentration of drug (or metabolite) in tumor tissue All cohorts except Cohort 6; target validation phase).

III. To assess changes in immune cell infiltration in DMG tumor tissue after 1 or 2 doses of ONC201 (All cohorts except Cohort 6; target validation phase).

IV. To assess correlation of intratumoral concentration of ONC201 with clinical outcome (All cohorts except Cohort 6; target validation phase).

V. To assess correlation of intratumoral drug concentration of novel agents with clinical outcome. (All cohorts except Cohort 6; target validation phase).

VI. To assess if intratumoral ONC201 concentrations differ in irradiated versus nonirradiated tumor tissue. (All cohorts except Cohort 6; target validation phase).

VII. To assess if intratumoral concentrations of novel agents differ in irradiated versus nonirradiated tumor tissue. (All cohorts except Cohort 6; target validation phase).

VIII. To assess tumor tissue biomarkers in the context of clinical outcome, such as PFS6 and/or OS12. (All cohorts except Cohort 6; target validation phase).

IX. To assess efficacy of combination therapy ONC201 and novel agent based on overall survival at 12 months (OS12). (All cohorts except Cohort 6; maintenance combinations).

X. To assess toxicity of combination therapy ONC201 and novel agents. (All cohorts except Cohort 6; maintenance combinations).

XI. To assess the toxicity of weekly ONC201 in combination with up-front radiation therapy. (Cohort 1; radiation therapy phase).

XII. To assess the toxicity of twice weekly ONC201 in combination with up-front radiation therapy. (Cohort 1; radiation therapy phase).

XIII. To assess the toxicity of novel agents in combination with up-front radiation therapy. (Cohort 1; radiation therapy phase).

XIV. To assess the toxicity of weekly ONC201 in combination with re-irradiation after progression. (Cohort 3).

XV. To assess the toxicity of twice weekly ONC201 in combination with re-irradiation therapy after progression. (Cohort 3).

XVI. To assess the toxicity of novel agents in combination with re-irradiation after progression. (Cohort 3).

XVII. To assess the toxicity of ONC201 in combination with novel agents in participants after re-irradiation after progression. (Cohort 3).

XVIII. To assess efficacy of a revised ONC201 dose and dosing schedule board based on median progression free survival (PFS) and overall survival (OS). (Cohort 4).

XIX. To assess efficacy of ONC201 in combination with targeted agent(s) that will be determined by a specialized tumor board based on median OS. (Cohort 5).

XX. To assess cerebrospinal fluid (CSF) biomarkers in the context of clinical outcome, such as PFS6 and/or OS12. (All cohorts except Cohort 6) XXI. To assess levels of circulating tumor deoxyribonucleic acid (ctDNA) in the context of imaging response criteria and clinical outcome, such as PFS6 and/or OS12. (All cohorts except Cohort 6) XXII. To assess single cell ribonucleic acid (RNA) sequencing in the context of clinical outcome, such as PFS6 and/or OS12. (All cohorts except Cohort 6) XXIII. To assess microbiome and flow cytometry studies in the context of imaging and clinical outcomes using descriptive statistics.(All cohorts except Cohort 6) XXIV. To assess Health-Related Quality of Life (HRQOL) and cognitive measures.(All cohorts except Cohort 6) XXV. To assess participants and/or proxy satisfaction with study participation via participant-reported outcome (PRO) measures. (All cohorts except Cohort 6) XXVI. To assess on therapy toxicity and survival in the context of race, ethnicity and other health related social risks. (All cohorts except Cohort 6) XXVII. To assess volumetric measurements of tumor in correlation with median OS. (All cohorts except Cohort 6) XXVIII. To assess MR spectroscopy of tumor in correlation with radiographic response, ONC201 exposure and median PFS and OS. (All cohorts except Cohort 6)

XXIX. To assess the therapeutic benefit including overall survival (OS), progression-free survival (PFS), the tumor objective response rate (ORR) and proportion of pseudoprogression (PSP) (Cohort 6) XXX. To assess the persistence of DNX-2401 antigen, DNA and transcripts in the tumor in the context of imaging response criteria and clinical outcome. (Cohort 6) XXXI. To assess the changes in cellular, molecular, and immunologic variables in the tumor in context of imaging response criteria and clinical outcome. (Cohort 6) XXXII. To assess the microbiome in the context of imaging response and clinical outcome. (Cohort 6) XXXIII. To assess peripheral blood biomarkers and cfDNA studies in the context of imaging and clinical outcome. (Cohort 6) XXXIV. To assess CSF biomarkers and cfDNA studies in the context of imaging and clinical outcomes. (Cohort 6) XXXV. To assess changes in functional status and in quality of life applying the PedsQLTM (Generic Score Scale). (Cohort 6) XXXVI. To assess patient and/or proxy satisfaction with study participation via patient-reported outcome (PRO) measures. (Cohort 6) XXXVII. To assess on therapy toxicity in the context of race, ethnicity and other health related social risks. (Cohort 6) XXXVIII. To assess volumetric measurements of tumor in correlation with median OS. (Cohort 6) XXXIX. To assess MR spectroscopy of tumor in correlation with radiographic response. (Cohort 6)

COHORT DESCRIPTIONS:

--ENROLLING-- COHORT 4A and 4B: Includes patients who are currently not eligible for defined combination arms of PNOC022 or other clinical trials investigating ONC201, such as ONC201-108 ACTION trial.

Cohort 4A^1: Includes newly diagnosed participants that have not yet undergone tumor tissue collection and have not yet completed radiation therapy.

Cohort 4A^2: Includes newly diagnosed participants that have not yet undergone tumor tissue collection and have completed radiation therapy. Cohort 4A^3: Includes participants with progressive DMG who are planned for SOC tumor collection and will undergo re-irradiation.

Cohort 4B^1: Includes newly diagnosed participants who have already undergone tumor tissue collection and have not yet completed radiation therapy.

Cohort 4B^2: Includes newly diagnosed participants who have already undergone tumor tissue collection and have completed radiation therapy. Cohort 4B^3: Includes participants with progressive DMG who are not planned for SOC tumor collection and will undergo re-irradiation.

--ENROLLING-- COHORT 5: Includes participants whose tumor demonstrates specific molecular alterations of interest considered targetable by an approved/available agent(s) and recommended by the PNOC022 tumor board. Participants are also allowed to receive ONC201 monotherapy with radiation or re-irradiation therapy.

Cohort 5^1: Includes newly diagnosed participants who have already undergone tumor tissue collection and have not yet completed radiation therapy.

Cohort 5^2: Includes newly diagnosed participants who have already undergone tumor tissue collection and have completed radiation therapy.

Cohort 5^3: Includes participants with progressive DMG who are not planned for SOC tumor collection and will undergo re-irradiation.

--ENROLLING-- COHORT 6: Includes participants with DMGs who have completed focal radiation therapy and are within 4-14 weeks from completion of radiation therapy without evidence of progression, who will undergo repeated intratumor DNX-2401 infusions.

-NOT CURRENTLY ENROLLING- COHORTS 1A & 2A (Target Validation cohorts); Includes newly diagnosed participants that have not yet undergone tumor tissue collection. Cohort 1A will include participants with DMG who have not yet completed radiation therapy and Cohort 2A will include participants with DMG who have completed radiation therapy.

-NOT CURRENTLY ENROLLING - COHORTS 1B & 2B: Includes newly-diagnosed participants who have already undergone tumor tissue collection. Cohort 1B will include participants with DMG who have not yet completed radiation therapy and Cohort 2B will include participants with DMG who have completed radiation therapy.

-NOT CURRENTLY ENROLLING- COHORTS 3A & 3B: Includes participants with progressive DMG. Cohort 3A will include participants planned for standard of care (SOC) tumor tissue collection. Cohort 3B will include participants not planned for SOC tumor tissue collection. The nomenclature will delineate participants previously enrolled in Cohorts 1 or 2.

-NOT CURRENTLY ENROLLING - COMBINATION COHORTS 1, 2 and 3: Participants are randomized to 1 of 3 arms.

ARM 2: During the trial validation phase, participants without prior biopsy receive ONC201 on day -1 prior to standard of care biopsy. During the radiation/re-irradiation phase, participants without prior radiation therapy or have disease progression after radiation therapy undergo weekly radiation therapy and receive ONC201 weekly during radiation therapy. During the maintenance phase, participants receive ONC201 weekly and paxalisib daily. Cycles repeat every 28 days (4 weeks) in the absence of adverse events of unacceptable toxicity.

ARM 4: During the trial validation phase, participants without prior biopsy receive ONC201 on days -2 and -1 prior to standard of care biopsy. During the radiation/re-irradiation phase, participants may receive ONC201 weekly during radiation therapy. During the maintenance phase, participants receive ONC201 weekly and paxalisib. Cycles repeat every 28 days (4 weeks) in the absence of adverse events or unacceptable toxicity.

ARM 6: During trial validation phase, participants without prior biopsy receive paxalisib on day -1 prior to standard of care biopsy. During the radiation/re-irradiation phase, participants without prior radiation therapy or have disease progression after radiation therapy undergo radiation therapy five times a week and receive paxalisib during radiation therapy. During the maintenance phase, participants receive ONC201 and paxalisib during each cycle. Cycles repeat every 28 days (4 weeks) in the absence of adverse events of unacceptable toxicity.

All Cohorts: After completion of study treatment, participants are followed at 30 days and then every 3 months for up to 5 years, until withdrawal of consent, or until death, whichever occurs first.

ELIGIBILITY:
--COHORTS 1, 2, AND 3 CLOSED---

INCLUSION CRITERIA:

COHORT 1A AND 1B:

* New diagnosis of DMG with imaging and/or pathology consistent with a DMG, including spinal cord tumors. In cohort 1B, previous tumor tissue confirmation of DMG is mandatory and pathology must be consistent with a DMG including diffuse midline glioma Histone 3 lysine 27 - mutant (H3K27M); World Health Organization (WHO) grade III and IV H3 wildtype gliomas.
* Must be within 6 weeks of diagnosis to begin standard of care radiation therapy on study.

COHORT 2A AND 2B:

* Diagnosis of DMG with imaging and/or pathology consistent with a DMG, including spinal cord tumors, who have complete standard-of-care radiation therapy. In Cohort 2B, previous tumor tissue confirmation of DMG is mandatory and pathology must be consistent with a DMG including diffuse midline glioma H3K27M mutant; WHO grade III and IV H3 wildtype gliomas.
* Participants must be within 4-14 weeks of completion of radiation. Radiation should have started within 6 weeks of diagnosis.

COHORT 3A AND 3B:

* Diagnosis of recurrent DMG with imaging and/or pathology consistent with a DMG, including spinal cord tumors, who have complete standard-of-care radiation therapy. In cohort 3B, previous tumor tissue confirmation of DMG is mandatory and pathology must be consistent with a DMG including diffuse midline glioma H3K27M mutant; WHO grade III and IV H3 wildtype gliomas.
* Participants must have evidence of progression and not have received any treatment for this progression and have not previously received re-irradiation.

COHORT 4A AND 4B:

* Diagnosis of DMG with imaging and/or pathology consistent with a DMG, including spinal cord tumors. In cohort 4B^1, previous tumor tissue confirmation of DMG is mandatory and pathology must be consistent with a DMG diffuse midline glioma H3K27-altered.
* Not currently eligible for any other clinical trials that include administration of ONC201.

Cohort 4A^1 and 4B^1 (participants with newly diagnosed DMG prior to radiation): Must be able to begin standard of care radiation therapy on study within 6 weeks of diagnosis.

Cohort 4A^2 and 4B^2 (participants with newly diagnosed DMG who have completed radiation): Participants must be within 4-14 weeks of completion of radiation and not have received additional therapy beyond completion of radiation therapy. Radiation should have started within 6 weeks of diagnosis.

Cohort 4A^3 and 4B^3 (participants with DMG at progression): Participants must have evidence of progression and not have received any treatment for this progression and have not previously received re-irradiation.

COHORT 5

* Diagnosis of DMG with imaging and/or pathology consistent with a DMG, including spinal cord tumors. In cohort 5^1, previous tumor tissue confirmation of DMG is mandatory and pathology must be consistent with a DMG diffuse midline glioma H3K27-altered.
* Not currently eligible for any other clinical trials that include administration of ONC201.
* Multifocal and leptomeningeal disease will be eligible for Cohort 5.
* Participant's tumor must demonstrate one of the following molecular alterations considered targetable by an approved agent:

  * BRAFV600E
  * PDGFRA (DNA point mutation or amplification with >=5 copy numbers)
  * FGFR1 (DNA point mutation, gene fusions, or amplification with >=5 copy numbers)
  * NF1

Cohort 5^1 (participants pre-radiation): Must be able to begin standard of care radiation therapy on study within 6 weeks of diagnosis.

Cohort 5^2 (participants post-radiation): Participants must be within 4-14 weeks of completion of radiation and not have received additional therapy beyond completion of radiation therapy. Radiation should have started within 6 weeks of diagnosis.

Cohort 5^3 (participants with progression): Participants must have evidence of progression and not have received any treatment for this progression and have not previously received re-irradiation.

All Cohorts (except Cohort 6):

* Age 2 to 39 years
* Participants must have recovered from all acute side effects of prior therapy and be beyond the window for expected ongoing acute toxicities. Any number of prior therapies are allowed.
* Prior ONC201 exposure is allowed, except in participants who have participated in Chimerix trials investigating ONC201 in the upfront setting. Participants who participated in trials investigating ONC201 in the upfront setting will not be eligible at any time, with the exception if participants received ONC201 as part of PNOC022 or other expanded access programs such as German sources of ONC201.
* Participant body weight must be above the minimum necessary for the participant to receive ONC201 (at least 10 kilograms (kg))
* From the projected start of scheduled study treatment, the following time periods must have elapsed: At least 7 days after last dose of a biologic agent or beyond time during which adverse events are known to occur for a biologic agent, 5 half-lives from any investigational agent, 4 weeks from cytotoxic therapy (except 23 days for temozolomide and 6 weeks from nitrosoureas), 6 weeks from antibodies (21 days for bevacizumab when used for tumor-directed therapy, guidance on use for pseudo-progression is below), or, or 4 weeks (or 5 half-lives, whichever is shorter) from other anti-tumor therapies.

  o The use of bevacizumab to control radiation therapy-induced edema is allowed (if used for tumor-directed therapy, please see required time period above).
  * Dosing limitations are as follows:
  * * Bevacizumab (or equivalent) for up to a maximum of 5 doses, dosing per institutional standard. There is no required washout period.
* Prior use of temozolomide during radiation at maximum of the standard pediatric dosing (defined as 90 mg/m2 /dose continuously during radiation therapy for 42 days) or dexamethasone is allowed. Any other agent given throughout radiation therapy must be discussed with the study chairs prior to beginning the agent.
* Corticosteroids: Participants who are receiving dexamethasone must be on a stable or decreasing dose for at least 3 days prior to baseline magnetic resonance imaging (MRI) scan.
* The participant must have adequate organ function defined as:

  * Peripheral absolute neutrophil count (ANC) >= 750/mm^3 (1.0g/l) AND
  * Platelet count >= 75,000/mm^3 (100x10^9/l) (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).
  * Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 OR
  * A serum creatinine within the normal limits for age
  * Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age AND
  * Serum glutamate pyruvate transaminase (SGPT)(alanine aminotransferase (ALT)) =< 3 x ULN AND
  * Serum albumin >= 2 g/Dl
  * No evidence of dyspnea at rest, no exercise intolerance due to pulmonary insufficiency, and a pulse oximetry of > 92% while breathing room air.
  * Diarrhea < grade 2 by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0
  * No history of congestive heart failure or family history of long QT syndrome.
  * ECG must be obtained to verify the Corrected QT Interval (QTc). If an abnormal reading is obtained, the ECG should be repeated in triplicate. QTC < 470 msec.
  * Participants with history of congestive heart failure, at risk of having or have underlying cardiovascular disease, or with history of exposure to cardiotoxic drugs must have adequate cardiac function as determined by echocardiogram. Shortening fraction of >= 27%.
  * Participants with seizure disorder may be enrolled if seizure disorder is well controlled
* Females of child-bearing potential and males must agree to use adequate contraception.
* Karnofsky >= 50 for participants > 16 years of age and Lansky >= 50 for participants =< 16 years of age. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Participants must be willing to provide adequate tissue. A minimum of 10-20 paraffin embedded unstained slides OR 1 block with tumor content of 40% or greater is required. Frozen tissue is also acceptable.

COHORT 6 Inclusion Criteria:

* Diagnosis of newly diagnosed thalamic or pontine located DMG with imaging and/or pathology consistent with a DMG, excluding spinal cord tumors, who have completed standard-of-care radiation therapy. If archival tissue is available prior to first biopsy, participants must be willing to provide adequate tissue. A minimum of 10-20 paraffin embedded unstained slides OR 1 block with tumor content of 40% or greater is required.
* Participants must be within 4-14 weeks of completion of radiation. Radiation should have started within 6 weeks of diagnosis.
* Age 2-39 years.
* Prior use of temozolomide during radiation at maximum of the standard pediatric dosing (defined as 90 mg/m2 /dose continuously during radiation therapy for 42 days) is allowed. Any other agent given throughout radiation therapy must be discussed with the study chairs prior to enrollment.
* Participants must have recovered from all acute side effects of prior therapy and be beyond the window for expected ongoing acute toxicities. Washout requirements from prior therapy include:

  * At least 7 days after last dose of a biologic agent or beyond time during which adverse events are known to occur for a biologic agent, 5 half-lives from any investigational agent, 4 weeks from cytotoxic therapy (except 30 days for temozolomide and 6 weeks from nitrosoureas), 6 weeks from antibodies (28 days for bevacizumab when used for tumor-directed therapy, guidance on use for pseudo-progression is below), or 4 weeks (or 5 half-lives, whichever is shorter) from other anti-tumor therapies.
  * At least 4 weeks prior to study enrollment from last immune therapy
* Corticosteroids: Participants treated with corticosteroids must be on stable or decreasing dose for at least 1 week prior to enrollment, with maximum dexamethasone dose 0.1 mg/kg/day dexamethasone equivalent at time of enrollment.
* The participant must have adequate organ function defined as:

  * Peripheral absolute neutrophil count (ANC) >= 750/mm3 (1.0g/l) and
  * Platelet count >= 75,000/mm3 (100x109/l) (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment.
  * Creatinine clearance or radioisotope GFR >= 70mL/min/1.73 m2 or
  * A serum creatinine within the normal limits for age.
  * Total bilirubin <= 3 x upper limit of normal (ULN); in presence of Gilbert's syndrome, total bilirubin </= 6 x ULN or direct bilirubin <= 3 x ULN
  * ALT <= 5 x ULN
  * AST <= 5 x ULN.
  * Serum albumin >= 2 g/dL
  * Diarrhea < grade 2 by CTCAE v5.0.
  * No history of congestive heart failure or family history of long QT syndrome.
  * Participants with seizure disorder may be enrolled if seizure disorder is well controlled.
* The effects of the study drugs on the developing human fetus are unknown. For this reason, females of child-bearing potential and males must agree to use adequate contraception.
* Karnofsky >/= 70 for Participants > 16 years of age and Lansky >/= 70 for participants </= 16 years of age. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score

EXCLUSION CRITERIA:

COHORT 1A AND 1B:

* Prior exposure to radiation therapy.
* Thalamic and Cerebellar H3K27M DMG.

COHORT 2A AND 2B:

* For tumors that do not have a pontine or spinal cord epicenter the following specific exclusion criteria apply:
* Thalamic and Cerebellar H3K27M DMG that has undergone standard radiation without concurrent therapy (other than temozolomide).

COHORT 1A AND 2A:

• Deemed not appropriate for tissue resection/biopsy.

COHORT 3A AND 3B:

* Prior exposure to re-irradiation for tumor progression.
* Thalamic and cerebellar H3K27M mutant DMG.

COHORT 4A AND 4B:

Cohort 4A^1and 4B^1: Prior exposure to radiation therapy Cohort 4A^3 and 4B^3: Prior exposure to re-irradiation for tumor progression

* Thalamic and cerebellar H3K27M mutant DMG, except those who received ONC201/ONC026 from alternative source prior to 2024 or US patients enrolled while the accelerated approval new drug application for dordaviprone to treat recurrent H3 K27M-mutant diffuse glioma is under review by US FDA.
* Cohort 4A^1and 4B^1: Prior exposure to radiation therapy
* Cohort 4A^3 and 4B^3: Prior exposure to re-irradiation for tumor progression

COHORT 5:

* Thalamic and cerebellar H3K27M mutant DMG, except those who received ONC201/ONC026 from alternative source prior to 2024 or US patients enrolled while the accelerated approval new drug application for dordaviprone to treat recurrent H3 K27M-mutant diffuse glioma is under review by US FDA.
* Cohort 5^1: Prior exposure to radiation therapy
* Cohort 5^3: Prior exposure to re-irradiation for tumor progression

All Cohorts (except Cohort 6):

* Diagnosis of a histone H3 wildtype grade II diffuse astrocytoma.
* Participants who are currently receiving another investigational drug. Investigational imaging agents or agents used to enhance tumor visibility on imaging or during tumor biopsy/resection should be discussed with the study chairs.
* Participants who are currently receiving other anti-cancer agents.
* Participants with a known disorder that affects their immune system, such as human immunodeficiency virus (HIV) or hepatitis B or C, or an auto-immune disorder requiring systemic cytotoxic or immunosuppressive therapy. Note: Participants that are currently using inhaled, intranasal, ocular, topical or other non-oral or non-intravenous (IV) steroids are not necessarily excluded from the study but need to be discussed with the study chair.
* Participants with uncontrolled infection or other uncontrolled systemic illness.
* Female participants of childbearing potential must not be pregnant or breast-feeding. Female participants of childbearing potential must have a negative serum or urine pregnancy test prior to the start of therapy (as clinically indicated).
* Active illicit drug use or diagnosis of alcoholism.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition as the agents used in study.
* Evidence of disseminated disease, including diffuse leptomeningeal disease or evidence of CSF dissemination, with the exception of Cohort 5.
* Known additional malignancy that is progressing or requires active treatment within 3 years of start of study drug.
* Concomitant use of potent CYP3A4/5 inhibitors during the treatment phase of the study and within 72 hours prior to starting study drug administration.
* Concomitant use of potent CYP3A4/5 inducers, which include enzyme inducing antiepileptic drugs (EIAEDs), during the treatment phase of the study and within 2 weeks prior to starting treatment. Concurrent corticosteroids is allowed.

COHORT 6 Exclusion Criteria:

* • DMGs located outside the thalamus and pons including bilateral thalamic tumors.
* Unacceptable anesthesia or surgery risk, as determined by the anesthesiologist or the neurosurgeon.
* Evidence of significant mass effect
* Evidence of herniation on imaging.
* Participants with a known history coagulopathy that increases risk of bleeding or a history of clinically significant hemorrhage within 12 months of registration.
* Participants must not require systemic anti-coagulation that cannot be halted for each intraoperative and perioperative biopsy time-period.
* Participants with active viral infection or who are currently receiving antiviral treatment.
* Participants with active, known, or suspected immunosuppressive disorders, such as acquired or congenital immune deficiency syndromes and autoimmune diseases.
* This virus infects cells with a deficit in the RB gene. Therefore, participants with Li-Fraumeni Syndrome or a known germ line deficit in the retinoblastoma gene or its related pathway are excluded.
* Participants must not have live or live-attenuated vaccinations within 30 days prior to DNX-2401 administration and while participating in the study. Killed vaccines are permitted.
* Participants who are currently receiving another investigational drug. Investigational imaging agents or agents used to enhance tumor visibility on imaging or during tumor biopsy/resection should be discussed with the study chairs.
* Participants with a known disorder that affects their immune system, such as HIV or Hepatitis B or C, or an auto-immune disorder requiring systemic cytotoxic or immunosuppressive therapy. Note: Participants who are currently using inhaled, intranasal, ocular, topical or other non-oral or non-IV steroids are not necessarily excluded from the study but need to be discussed with the study chair(s).
* Participants with uncontrolled infection or other uncontrolled systemic illness.
* Female participants of childbearing potential must not be pregnant or breast-feeding. Female participants of childbearing potential must have a negative serum or urine pregnancy test prior to the start of therapy (as clinically indicated).
* Active illicit drug use or diagnosis of alcoholism.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition as the agents used in the study.
* Evidence of disseminated disease, including multi-focal disease, diffuse leptomeningeal disease or CSF dissemination.

Ages: 2 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival at 6 months (PFS6) - Cohorts 1A, 1B Only | 6 months after diagnosis
  Percentage of participants alive and free from progression at 6 months after the diagnosis. The primary analysis for PFS6 is based on the intention to treat (ITT) population, according to treatment arm assignment. PFS6 is estimated using the Kaplan-Meier method with exact confidence intervals for each cohort and arm. Participants with unknown progression status at 6 months are considered failures (i.e., progressed) for the PFS6 analysis.
Progression-free survival at 6 months (PFS6) - Cohorts 2A, 2B Only | 6 months after diagnosis
  Percentage of participants alive and free from progression at 6 months after diagnosis. The primary analysis for PFS6 is based on the intention to treat (ITT) population, according to treatment arm assignment. PFS6 is estimated using the Kaplan-Meier method with exact confidence intervals for each cohort and arm. Participants with unknown progression status at 6 months are considered failures (i.e., progressed) for the PFS6 analysis.
Overall survival at 7 months (OS7) - Cohort 3A & 3B Only | 7 months after administration of ONC201 in the maintenance phase
  OS7 is defined as the percentage of participants alive at 7 months after the initiation of the combination of the backbone (i.e., ONC201) with a novel agent given in the maintenance phase of therapy. The primary analysis for OS7 is based on the ITT population, according to treatment arm assignment. OS7 is estimated using the Kaplan-Meier method with exact confidence intervals for each cohort and arm. Participants with unknown survival status at 7 months are considered failures (i.e., dead) for the OS7 analysis.
Proportion of participants reporting dose-limiting toxicities (DLTs) (Cohort 4) | Up through the first cycle of maintenance therapy, approximately 8 months
  The safety and tolerability of ONC201 at a previously untested dose will be measured by the proportion of participants reporting a DLT within the first cycle of treatment.
Number of participants requiring dose modification through first cycle of maintenance (Cohort 5) | Up through the first cycle of maintenance therapy, approximately 8 months
  The safety and tolerability of ONC201 in combination with targeted therapies will be measured by the number of participants reporting dose modification during first cycle.
Maximum tolerated number of intratumor infusions of DNX-2401, with a maximum of 6, in participants with thalamic or pontine DMG who have completed radiotherapy (Cohort 6) | A maximum of 6 infusions will be administered every 30 days - approximately 8 months
  The safety and tolerability of DNX-2401 at Dose Level 1 (5 × 10^10 viral particles) will be measured by the proportion of participants reporting a DLT.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (32):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, San Diego / Rady Children's Hospital, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Children's National Hospital, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University Riley Children's Hospital, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Dana-Farber Cancer Institute Harvard University, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospital Minnesota, Minneapolis, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Hackensack Meridian Health, Hackensack, New Jersey
  - New York University, New York, New York
  - Duke University, Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Australia (8):
  - John Hunter Children's Hospital, New Lambton Heights, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Monash Children's Hospital, Clayton, Victoria
  - The Royal Children's Hospital Melbourne, Melbourne, Victoria
  - Perth Children's Hospital, Nedlands, Washington
  - Women and Children's Hospital, Adelaide
  - Sydney Children's Hospital, Sydney
- Israel (2):
  - Sheba Medical Center, Tel Litwinsky, Ramat Gan
  - Shaare Zedek Medical Center, Jerusalem
- Princess Maxima Center, Utrecht, Netherlands
- Starship Children's Hospital, Auckland, New Zealand
- The University Children's Hospital in Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data after de-identification will be shared with study collaborators
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Jackson ER, Duchatel RJ, Staudt DE, Persson ML, Mannan A, Yadavilli S, Parackal S, Game S, Chong WC, Jayasekara WSN, Grand ML, Kearney PS, Douglas AM, Findlay IJ, Germon ZP, McEwen HP, Beitaki TS, Patabendige A, Skerrett-Byrne DA, Nixon B, Smith ND, Day B, Manoharan N, Nagabushan S, Hansford JR, Govender D, McCowage GB, Firestein R, Howlett M, Endersby R, Gottardo NG, Alvaro F, Waszak SM, Larsen MR, Colino-Sanguino Y, Valdes-Mora F, Rakotomalala A, Meignan S, Pasquier E, Andre N, Hulleman E, Eisenstat DD, Vitanza NA, Nazarian J, Koschmann C, Mueller S, Cain JE, Dun MD. ONC201 in Combination with Paxalisib for the Treatment of H3K27-Altered Diffuse Midline Glioma. Cancer Res. 2023 May 17:OF1-OF17. doi: 10.1158/0008-5472.CAN-23-0186. Online ahead of print. PMID 37195023
- [Derived] Jackson ER, Duchatel RJ, Staudt DE, Persson ML, Mannan A, Yadavilli S, Parackal S, Game S, Chong WC, Jayasekara WSN, Le Grand M, Kearney PS, Douglas AM, Findlay IJ, Germon ZP, McEwen HP, Beitaki TS, Patabendige A, Skerrett-Byrne DA, Nixon B, Smith ND, Day B, Manoharan N, Nagabushan S, Hansford JR, Govender D, McCowage GB, Firestein R, Howlett M, Endersby R, Gottardo NG, Alvaro F, Waszak SM, Larsen MR, Colino-Sanguino Y, Valdes-Mora F, Rakotomalala A, Meignan S, Pasquier E, Andre N, Hulleman E, Eisenstat DD, Vitanza NA, Nazarian J, Koschmann C, Mueller S, Cain JE, Dun MD. ONC201 in combination with paxalisib for the treatment of H3K27-altered diffuse midline glioma. Cancer Res. 2023 May 5;83(14):2421-37. doi: 10.1158/0008-5472.CAN-23-0186. Online ahead of print. PMID 37145169
- [Derived] Przystal JM, Cianciolo Cosentino C, Yadavilli S, Zhang J, Laternser S, Bonner ER, Prasad R, Dawood AA, Lobeto N, Chin Chong W, Biery MC, Myers C, Olson JM, Panditharatna E, Kritzer B, Mourabit S, Vitanza NA, Filbin MG, de Iuliis GN, Dun MD, Koschmann C, Cain JE, Grotzer MA, Waszak SM, Mueller S, Nazarian J. Imipridones affect tumor bioenergetics and promote cell lineage differentiation in diffuse midline gliomas. Neuro Oncol. 2022 Sep 1;24(9):1438-1451. doi: 10.1093/neuonc/noac041. PMID 35157764